CLINICAL TRIAL: NCT02022176
Title: Dietary Inorganic Nitrate: Effects on Metabolic Rate, Reactive Oxygen Species Production, Glucose Uptake and Primary Myotube Respiration.
Brief Title: Modulation of Metabolic Rate by Inorganic Nitrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Eddie Weitzberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JETF-6996-NO
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Resting Metabolic Rate
Keywords: Nitrate; Nitrite; Nitric oxide; Resting metabolic rate; Glucose uptake; Insulin sensitivity; Reactive oxygen species production; inorganic nitrate; Sodium nitrite infusion
MeSH Terms: conditions — Insulin Resistance | interventions — Basal Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Sodium nitrate (Active Comparator): 0.1 mmol NaNO3 / kg bodyweight / day for three days.
  Interventions: Other: Glucose Uptake; Other: Resting metabolic rate
- Sodium Chloride (Placebo Comparator): 0.1 mmol NaCl / kg bodyweight / day for three days.
  Interventions: Other: Glucose Uptake; Other: Resting metabolic rate
- Sodium nitrite infusion (Active Comparator): Sodium nitrite (NaNO2) at a rate of 1, 10 and 100 nmol kg-1 min-1 (10 minutes per dose) was infused intravenously.
  Interventions: Other: Nitrite infusion
- Saline infusion (Placebo Comparator): Saline at a rate corresponding to 1, 10 and 100 nmol NaCl kg-1 min-1 (10 minutes per dose) was infused intravenously.
  Interventions: Other: Nitrite infusion

INTERVENTIONS:
Other: Glucose Uptake — Glucose uptake is measured by oral glucose tolerance test and euglycemic clamp
  Arms: Sodium Chloride; Sodium nitrate
Other: Resting metabolic rate — Resting metabolic rate is measured by indirect calorimetry after an over-night fast
  Arms: Sodium Chloride; Sodium nitrate
Other: Nitrite infusion — Sodium nitrite or saline was infused at escalating doses at a rate of 1, 10 or 100 nmol kg-1 min-1 (10 minutes per dose) in a randomized, double blinded cross-over fashion
  Arms: Saline infusion; Sodium nitrite infusion

SUMMARY:
The purpose of this study is to determine the effects of sodium nitrate on resting metabolic rate, glucose uptake and formation of reactive oxygen species in humans.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

Exclusion Criteria Chronic medication Vegetarian Nicotine Users Known metabolic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate | day 4
  Resting metabolic rate, measured after overnight fast using indirect calorimetry

SECONDARY OUTCOMES:
Thyroid hormone status | day 4
Glucose uptake | day 4
  Glucose uptake measured with oral glucose tolerance test and euglycemic clamp
Nitrite infusion | 30 minutes
  Effect on resting metabolic rate when infusing escalating intravenous doses of sodium nitrite or saline solution

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Larsen FJ, Schiffer TA, Borniquel S, Sahlin K, Ekblom B, Lundberg JO, Weitzberg E. Dietary inorganic nitrate improves mitochondrial efficiency in humans. Cell Metab. 2011 Feb 2;13(2):149-59. doi: 10.1016/j.cmet.2011.01.004. PMID 21284982